CLINICAL TRIAL: NCT03730064
Title: Neuroinflammation as a Novel Target to Treat Bipolar Depression: A Pilot PET Study With [11C]PBR-28 and N-Acetyl Cysteine (NAC) Antidepressant Treatment
Brief Title: Brain Imaging to Understand the Role of Inflammation in N-Acetyl Cysteine (NAC) Treatment of Bipolar Depression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Martin Lan (Other)
Responsible Party: Sponsor-Investigator, Martin Lan, Assistant Professor of Psychiatry, New York State Psychiatric Institute
Organization: New York State Psychiatric Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7580
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Bipolar Disorder; Depression
Keywords: Inflammation; NAC; N-acetyl cysteine
MeSH Terms: conditions — Bipolar Disorder; Depression; Inflammation | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bipolar depressed (Experimental)
  Interventions: Drug: N-acetyl cysteine (NAC)

INTERVENTIONS:
Drug: N-acetyl cysteine (NAC) — Experimental medication with N-acetyl cysteine (NAC) for six weeks

SUMMARY:
We are trying to understand what causes bipolar disorder and how medications treat bipolar depression. Particularly, we are looking at the importance of inflammation in the process. If you participate, you will have two different brain scans (MRI and PET scan). You will also have an experimental treatment for your depression named N-acetyl cysteine (NAC). The study is funded by the Columbia University Irving Institute to improve the treatment of bipolar disorder. Please contact us if you are interested in participating. Up to $600 in compensation if you are eligible and choose to participate. Up to 6 months of treatment for depression at no cost to you.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar 2 disorder and meets criteria for a major depressive episode
* Age 18-60
* Females of child-bearing potential must be willing to use an acceptable method of birth control throughout the study
* Not currently taking psychotropic medications besides those allowed in the clinical trial

Exclusion Criteria:

* Failed trial or intolerable side effects of NAC
* Diagnosis of other major psychiatric disorders such as lifetime schizophrenia, schizoaffective disorder, psychotic features of bipolar disorder, current drug or alcohol abuse or recent drug or alcohol dependence
* Significant active physical illness, including blood dyscrasias, lymphomas, hypersplenism, endocrinopathies, renal failure, chronic obstructive lung disease, autonomic neuropathies, peripheral vascular disease. Any disorders with inflammation, malignancy, autoimmune or infectious etiology. Systolic blood pressure >140 or diastolic blood pressure > 100 Hemoglobin <11 in females or <13 in males
* Metal implants, pacemaker, metal prostheses, metal orthodontic appliances or shrapnel in the body
* Current, past or anticipated exposure to radiation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | Six weeks
  Total score will be used; Ranges from 0 to 60 points; 60 is more most severe depression

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No